CLINICAL TRIAL: NCT05911074
Title: Performance Assessment of COVID-19 Antigen Rapid Diagnostic Tests and Algorithms in Low-Prevalence Settings
Brief Title: COVID-19 Antigen Rapid Test Evaluation in Low-Prevalence Setting
Acronym: CV006
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other)
Responsible Party: Sponsor
Other Study IDs: CV006
Record Dates: First submitted 2023-06-19; First posted 2023-06-20 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Corona Virus Infection
Keywords: Covid 19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The SD Biosensor COVID-19 Ag test kit: This is one of the Investigational product or medical device(s) intended to be used with a study participant according to the study protocol
  Interventions: Diagnostic Test: The Abbott Panbio™ COVID-19 Ag Rapid Test

INTERVENTIONS:
Diagnostic Test: The Abbott Panbio™ COVID-19 Ag Rapid Test — This is the intervention or medical device(s) intended to be used with a study participant according to the study protocol.

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the resulting COVID-19 pandemic present important diagnostic challenges. Point-of-care tests that detect SARS-CoV-2 antigen have the potential to allow earlier detection and isolation of confirmed cases compared to PCR-based diagnostic methods, and could be implemented at Ports of Entry (PoE) to screen low-prevalence populations effectively.This study will assess the performance of available antigen Ag-RDTs such as the Panbio and Standard Q SARS-CoV-2 rapid antigen tests. Approximately 15,000 subjects entering Botswana at Ports of Entry will be enrolled over a 6-months period or more. SARS-CoV-2 RT-PCR will be used as a reference standard. A subset of participants will also be contacted, re-evaluated and re-tested at 48-72 hours following initial assessment, to assess for the impact of incubating infection on the performance of the Ag-RDTs.

In order to assess the impact of viral genetic variability on test performance, genomic sequencing will be part of the study. All SARS-CoV-2 PCR positive samples will undergo genomic sequencing to determine the virus lineages or variants.

In addition to assessing the performance of each of the Ag-RDTs, a set of testingalgorithms that could be implemented at Ports of Entry, including the sequential use of multiple Ag-RDTs with or without RT-PCR confirmation, will be assessed.

DETAILED DESCRIPTION:
Point-of-care tests to detect active SARS-CoV-2 infection have the potential to allow earlier detection and isolation of confirmed cases compared to PCR-based diagnostic methods performed in centralized laboratories, with the aim of cost-effective reduction of transmission field (Dinnes et al., 2020). In theory, sufficiently sensitive and specific point-of-care format tests could be implemented at PoE and used to screen low-prevalence populations effectively.

In particular, rapid COVID-19 antigen tests in a lateral flow format COVID antigen RDTs or AgRDTs can play a key role in accelerating access to testing and improving turnaround times for COVID-19 test results. COVID antigen RDTs detect specific proteins known as antigens on the surface of the virus and can identify people who are at the peak of infection when virus levels in the body are likely to be high. A number of AgRDTs are now available, some of which have received emergency use authorizations from the World Health Organisation (WHO) and/or the United States Food and Drug Administration (FDA). These tests have the potential to detect an active infection with performance that is close to that of PCR in specific settings. However, the performance of COVID antigen RDTs outside of highly controlled settings is not well defined,particularly in low-prevalence groups of asymptomatic people (Bryan et al., 2020; Lassaunière et al., 2020 Linares et al., 2020; Porte et al., 2020).

Antigen tests with rapid turnaround times and minimal user skill have been recently approved for emergency use listing (EUL) by the WHO. Performance data show sensitivity and specificity levels (at least 80% and 97%, respectively) sufficient for diagnostic purposes of SARS-CoV-2 in targeted individuals, but their role in population-based screening remains to be established. In this evaluation, performance characteristics of rapid SARS-COV-2 detection kits (including but not limited to the Standard Q COVID-19 Antigen Test Standard Q RDT and the Panbio™ COVID-19 Ag Rapid Test Panbio RDT, will be assessed for sensitivity, specificity, and their overall agreement with standard nucleic acid testing using polymerase chain reaction (PCR) tests. Finally, the performance of multi-test algorithms based on Ag-RDTs with or without RTPCR will be assessed for their potential use in low-prevalence screening programmes.

ELIGIBILITY:
Inclusion Criteria:

* In order to meet the study objectives, study recruitment will focus on the population meeting the following eligibility criteria:
* Age ≥ 18 years crossing ports of entry in Greater Gaborone Health District [including International Airport, Ports within Gaborone Health Districts ((as above)
* Able to understand the scope of the study and provided written informed consent

Exclusion Criteria:

* Participants are excluded from the study if any of the following exclusion criteria apply:
* Participants who are less than 18 years or who are unable to provide informed consent.
* Any contraindications to nasopharyngeal sample collection: recent nasal trauma or surgery, markedly deviated nasal septum, or a history of chronically blocked nasal passages or severe coagulopathy
* Vulnerable populations as deemed inappropriate for study by site PI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both male and female
Study Population: Study participants will be enrolled at PoE at study sites within the Greater Gaborone Health District.
  1. Sir Seretse Khama International Airport
  2. Tlokweng, Ramotswa, Pioneer and Ramatlabana land borders Participants will be included regardless of symptoms. Individuals younger than 18 years of age or unable to provide informed consent will be excluded from the study. A subset of study subjects are expected to show evidence of negative SARS-CoV-2 RT-PCR testing within the 72 hours prior to study enrolment. These subjects will be eligible for the study; however, based on the sample size considerations described above, the number of subjects with documented negative RT-PCR testing will be capped at 1,000.
Sampling Method: Non-Probability Sample
Enrollment: 7274 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Performance characteristics of two currently available Ag-RDTs for the detection of SARS-CoV-2 antigens in nasal swabs | 6 months
  Point estimates of sensitivity and specificity of the COVID-19 antigen RDTs compared to the reference standard reverse transcription polymerase chain reaction when used at ports of entry

SECONDARY OUTCOMES:
Cost estimates of Ag testing compared to PCR testing for COVID-19 case detection | 6 months
  (1) Cost per test performed for each of the Ag RDTs compared to RT-PCR based protocols
  (1) Cost per COVID-19 case detected for each of the Ag RDTs compared to RT-PCR based protocols

CONTACTS AND LOCATIONS:
Overall Officials: Sikulile Moyo, Phd, Principal Investigator — Botswana Harvard Aids Initiative Partneship
Locations (1):
- Botswana Harvard AIDS Institute Partnership, Gaborone, Gabonone, Botswana

IPD SHARING:
Plan to Share IPD: No
All manuscripts reporting FIND study data and all review articles with FIND authors should be published in an open-access, peer-reviewed journal, regardless of whether they are FIND-led or partner-led

REFERENCES:
- [Result] Hussong D, Damare JM, Limpert RJ, Sladen WJ, Weiner RM, Colwell RR. Microbial impact of Canada geese (Branta canadensis) and whistling swans (Cygnus columbianus columbianus) on aquatic ecosystems. Appl Environ Microbiol. 1979 Jan;37(1):14-20. doi: 10.1128/aem.37.1.14-20.1979. PMID 104659